CLINICAL TRIAL: NCT04828460
Title: Monitoring of COVID-19 Vaccine Response in Organ Transplant Patients
Acronym: COVATRANS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8133
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Kidney Transplantation
Keywords: covid19; kidney transplantation; seroconversion; immunosuppression; vaccination
MeSH Terms: conditions — COVID-19; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipients who receive Covid-19 vaccine

SUMMARY:
Vaccination against SARS CoV-2 appears to be the best strategy today to control the COVID-19 pandemic. The first published studies with Pfizer, Moderna and Astra-Zeneca vaccines show very good vaccine protection in the general population and good short-term tolerance. The efficacy of these vaccines ranges from 62 to 95%, which is particularly remarkable, especially for mRNA vaccines. Nevertheless, these studies do not report the vaccine response in organ transplant patients.

It is known that transplant patients have lower vaccine responses than immunocompetent patients due to some degree of immunosuppression.

Therefore, the investigators are interested in evaluating the vaccine response of organ transplant recipients after vaccination against SARS- CoV-2. For non-responder patients, new strategies can be proposed: 3rd or 4th boost of vaccine or perfusion/injection of antiS monoclonal antibodies. These strategies must be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, adult or child (15 years and older)
* Patient vaccinated against SARS-CoV-2 as part of routine care, and having received the 2 injections
* Solid organ transplant recipient
* Transplantation for more than 3 months

Exclusion Criteria:

* History of anaphylactic shock or known allergy to PEG
* Known history of COVID or positive Covid serology in the 3 months preceding inclusion
* Formal contraindication to an intra-muscular injection
* Impossibility to give the subject informed information (subject in emergency situation, difficulties in understanding the subject, ...)
* Subject under legal protection
* Subject under guardianship or curatorship
* Patient having expressed his opposition to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients followed in French transplant centers
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who develop a seroconversion for SARS Cov-2 anti Spike antibodies | One month after the 2nd injection of the COVID-19 vaccine

SECONDARY OUTCOMES:
Compare the seroconversion between different vaccines | At Month 3, Month 6, Month12 and Month 24 after the 2nd injection of the COVID-19 vaccine
Percentage of patients who develop a seroconversion for SARS Cov-2 anti Spike antibodies | At Month 3, Month 6, Month12 and Month 24 after the 2nd injection of the COVID-19 vaccine and at Month 1 after the 3rd and 4th injection.
Describe the patients characteristics associated with seroconversion | At Month 24 after the 2nd injection of the COVID-19 vaccine
Assess the tolerance of the 3rd and 4th doses of vaccine in transplant patients | At the day of injection, Month 1, Month 2, Month 3, Month 6 and Month 12 post injection
Percentage of patients who develop a Seroconversion for SARS Cov-2 anti Spike and anti N antibodies after injection of monoclonal antibodies | At Month 1, Week 6, Week 8, Month 3, Month 6 and Month 12 afin injection of monoclonal antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France